CLINICAL TRIAL: NCT04680533
Title: Transcutaneous Electrical Nerve Stimulation for Peripheral Edema: A Single Arm Clinical Trial
Brief Title: Wireless TENS for Peripheral Edema (Lower Limb Swelling)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Terminated early due to lack of time.
Sponsor: University of Rochester (Other)
Collaborators: NeuroMetrix, Inc. (Industry)
Responsible Party: Principal Investigator, Jennifer Gewandter, Assistant Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005655
Record Dates: First submitted 2020-12-10; First posted 2020-12-23 (Actual); Results first posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Peripheral Edema
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Single Arm
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- TENS device (Experimental): The device is worn on the upper calf right below the knee and secured by an elastic band. The device is controlled by an App and alternates between treatment periods and rest periods. Participants will be asked to wear the device 7-8 hours per day alternating legs.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS)

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation (TENS) — Quell TENS device. The device is worn on the upper calf right below the knee and secured by an elastic band. The device is controlled by an App and alternates between treatment periods and rest periods. Participants will be asked to wear the device 7-8 hours per day alternating legs.

SUMMARY:
This study is single center, subject will receive a wireless TENS device. All subjects will be allowed to keep the commercially-available device for use after the study. The primary goal is to test the feasibility of the study design and secondary is to test the preliminary efficacy of the TENS.

DETAILED DESCRIPTION:
This study is single center, subject will receive a wireless TENS device. The coordinator will introduce the study device, be available to answer questions about the device, and assess adverse events. Subjects will be told that we are testing whether TENS, which has shown promise in some patients but needs to be tested formally, has an effects on lower limb swelling . The treatment period will be 3 weeks in duration. After the treatment period, all subjects will be asked to complete the Treatment-period Endpoint-Qualitative interview. All subjects will be allowed to keep the commercially-available device for use after the study.

ELIGIBILITY:
Inclusion criteria (subjects must…)

1. Have had lower extremity edema for at least 3 months.
2. Currently have edema of at least 2+ (i.e., 3-4mm depression rebounds within a few seconds, but not immediately) on the pitting scale. 21 Pitting will have been assessed by a Clinician, the clinician Co-I within 6 weeks of the screening visit or at the screening visit by the research staff.
3. Willing to not start or change the dosages of any medications that could affect edema for 2 weeks prior to enrollment, and throughout the duration of the study.
4. Not currently using diuretics to control their edema.
5. Not currently using and willing to not start using occupational therapy, physical therapy, or lymphatic massage (at home or by PT) 2 weeks prior to and throughout the duration of the study.
6. Not currently using compression stockings or Velcro or bandage wraps at least 2 weeks prior to enrollment in the study or based on shared decision making of the potential subjects' clinician or the clinician co-investigator are receiving sufficiently little benefit from these therapies to warrant stopping their use for the duration of the study.
7. Have access to a smart phone or device with an Apple or Android operating system with iOS 10 or later, or Android 6 or later. iOS and Android devices must have Bluetooth Low Energy (LE, also called Bluetooth Smart) compatibility. The smart phone or device must have the ability to access the TENS device's Quell App, Zoom App or software and, the ability to connect to the cellular data or Wi-Fi on a daily basis during the trial.
8. Have an active and accessible email.
9. Be willing and able to regularly check the email provided throughout the study.
10. Be able to read English (i.e., is literate, can speak English, and is not blind) because patient-reported outcomes and consent form are only available in English.
11. Be at least 18 years of age.
12. Be able to provide informed consent.

Exclusion criteria (subjects must not…)

1. Be currently using a TENS device for any reason.
2. Have an acute and symptomatic lower extremity DVT (i.e., the diagnosis of DVT is less than 3 months prior to study enrollment).
3. Have started anticoagulants within the past 3 months.
4. Have lower extremity wounds or ulcers.
5. Have a cardiac pace maker or defibrillator.
6. Have epilepsy.
7. Have a leg that is too small or too large for the TENS device to fit securely.
8. Have cellulitis or fibrosis.
9. Have any skin condition at the site where the electrode pads adhere such that the PI/Co-I think the device will not be safe for the subject.
10. Have congestive heart failure.
11. Have chronic kidney disease of stage 3 or greater.
12. Have cirrhosis of the liver.
13. Have previous surgery that removed lymphatic lower leg tissue.
14. Have a diagnosis of lower limb lymphedema.
15. Be pregnant or planning to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-02-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TENS device
Started | 3
Completed | 2
Not Completed | 1
Not completed — Screen failure | 1

BASELINE CHARACTERISTICS:
Arm/Group | TENS Device
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants] — Population: One subject did not answer the question, so only 2 responses were entered out of 3 subjects.
  Participants
    number analyzed (Participants) | 2
    <=18 years | 0
    Between 18 and 65 years | 1
    >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Edema Symptom Diary Score
Description: Swelling and symptoms associated with edema will be recorded in the Edema Symptom Diary using a verbal rating scale of swelling in the lower limbs and feet using the anchors "none", "a little bit", "quite a bit" "a lot", or "very much", which converts to a 1 to 5 measurable scale, with [1 = none, 5 = very much]. The scores per each symptom per day will be summed and averaged over 7 days. The higher the score the worse the health outcome. The range of scores the participant can achieve per day is between 6 - 30.
Time Frame: From baseline visit (Day 0) to final endpoint visit (Day 21)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TENS device
Number analyzed (Participants) | 2
score on a scale | -5.5 (1.5)

2. Secondary Outcome: Mean Change in Coordinator Tape Measurements of the Lower Limb
Description: The blinded coordinator measures the arch of the foot, the midpoint between the kneecap and ankle, and the knee crease on both limbs, regardless of which is more affected. These measurements are recorded in the Coordinator Lower Limb Swelling form. For analysis, the individual measurements are summed for each visit, and the average of these sums across relevant records is calculated separately for baseline and final endpoint visits to assess changes over time.
Time Frame: From baseline visit (Day 0) to final endpoint visit (Day 21)
Measure: Mean (Standard Deviation); unit: CM
Units Other Than Participants: lower limbs
Arm/Group | TENS device
Number analyzed (Participants) | 2
Number analyzed (lower limbs) | 2
CM
  Mean Baseline | 236.5 (9.5)
  Mean Final Endpoint | 230.6 (0)

3. Secondary Outcome: Mean Change in Patient Global Impression of Change in Edema Symptoms Score
Description: The Patient Global Impression of Change in Edema Symptoms (PGIC-Edema) form contains multiple items, each rated on a 1-7 scale, with 1 = "very much improved," 4 = "not changed," and 7 = "very much worse." The total score is the sum of all item scores, with a possible range of 0-105. Higher scores indicate worse edema symptoms. For each participant, the baseline total score and final endpoint total score (Day 21) were calculated, and mean change was defined as the value at the final endpoint visit minus the value at the baseline visit.
Time Frame: Baseline visit (Day 0) and final endpoint visit (Day 21)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TENS device
Number analyzed (Participants) | 2
score on a scale | 53 (6)

4. Secondary Outcome: Mean Change in Lymphoedema Quality of Life Questionnaire (LYMQOL) Score
Description: The Lymphoedema Quality of Life Questionnaire (LYMQOL) contains 26 items, each scored on a 0-4 scale, where 0 = "not at all" and 4 = "very much." Higher scores indicate worse quality of life. The total score is the sum of all item scores, with a possible range of 0-104. For each participant, the baseline total score and final endpoint total score (Day 21) were calculated, and mean change was defined as the value at the final endpoint visit minus the value at the baseline visit.
Time Frame: Baseline visit (Day 0) and final endpoint visit (Day 21)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TENS device
Number analyzed (Participants) | 2
score on a scale
  Mean Baseline | 36 (2)
  Mean Final Endpoint | 38 (11)

ADVERSE EVENTS:
Time Frame: from enrollment until end of follow-up, up to 2 months
Arm/Group | TENS device
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 1/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TENS device (N=3)
contact dermatitis (Skin and subcutaneous tissue disorders) | 1
Vertigo (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-06): https://cdn.clinicaltrials.gov/large-docs/33/NCT04680533/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/33/NCT04680533/ICF_001.pdf